CLINICAL TRIAL: NCT01734850
Title: An Adaptive Phase I/II Study of the Safety of CD4+ T Lymphocytes and CD34+ Hematopoietic Stem/Progenitor Cells Transduced With LVsh5/C46, a Dual Anti-HIV Gene Transfer Construct, With and Without Conditioning With Busulfan in HIV-1 Infected Adults Previously Exposed to ART
Brief Title: Safety Study of a Dual Anti-HIV Gene Transfer Construct to Treat HIV-1 Infection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Calimmune, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CAL-USA-11
Record Dates: First submitted 2012-11-19; First posted 2012-11-28 (Estimated); Results first posted 2020-08-06 (Actual); Last update posted 2020-08-06 (Actual); Status verified 2020-07

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV-1
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Busulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No busulfan pre-conditioning (Experimental): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes without busulfan preconditioning
  Interventions: Biological: Cal-1 modified HSPC; Biological: Cal-1 modified CD4+ T lymphocytes
- 1 x 4mg/kg busulfan preconditioning (Experimental): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes, with single 4mg/kg busulfan dose administered as pre-conditioning for transplant
  Interventions: Drug: Busulfan; Biological: Cal-1 modified HSPC; Biological: Cal-1 modified CD4+ T lymphocytes
- 2 x 4mg/kg busulfan pre-conditioning (Experimental): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes, with two 4mg/kg busulfan doses administered as pre-conditioning for transplant
  Interventions: Drug: Busulfan; Biological: Cal-1 modified HSPC; Biological: Cal-1 modified CD4+ T lymphocytes

INTERVENTIONS:
Drug: Busulfan — Intravenous busulfan
  Other Names: Busulfex
  Arms: 1 x 4mg/kg busulfan preconditioning; 2 x 4mg/kg busulfan pre-conditioning
Biological: Cal-1 modified HSPC — Hematopoietic progenitor/stem cells (HSPC) modified with LVsh5/C46 (Cal-1)
  Other Names: LVsh5/C46 modified HSPC
Biological: Cal-1 modified CD4+ T lymphocytes — CD4+ T lymphocytes modified with LVsh5/C46 (Cal-1)
  Other Names: LVsh5/C46 modified CD4+ T lymphocytes

SUMMARY:
This is an early phase research study looking at whether an experimental gene transfer, LVsh5/C46 (also known as Cal-1), is safe and if it can protect the immune system from the effects of HIV without the use of antiretroviral drugs.

Cal-1 is an experimental gene transfer agent designed to inhibit HIV infection through 2 active parts:

1. Removing a protein named CCR5 from bone marrow and white blood cells
2. Producing a protein named C46 on bone marrow and white blood cells

DETAILED DESCRIPTION:
It is estimated that 33 million individuals are currently infected with HIV. HIV/AIDS is a disease that impairs immune function, primarily by decreasing CD4+ T lymphocytes. The progression can be contained by daily dosing with antiretroviral therapy (ART) but there are side effects that can be treatment limiting, and the development of HIV drug resistance can force the physician to modify the ART regimen. There are no effective vaccines currently available for HIV.

LVsh5/C46 (also known as Cal-1) is a dual therapeutic, self-inactivating lentiviral vector that encodes for both a short hairpin RNA against the HIV-1 co-receptor CCR5 (sh5) and a HIV-1 fusion inhibitor, C46 and inhibits two processes required for HIV-1 infection:

1. Binding of the virus to the cellular CCR5 co-receptor and
2. Fusion of the virus with the host cell

The rationale is that Cal-1 introduced into hematopoietic progenitor/stem cells (HSPC) and mature CD4+ T lymphocytes will protect these cells and their progeny cells from HIV-1 infection and its pathogenic sequelae. This may provide a continuous means of controlling HIV-1 after a single or infrequent dose(s), thereby decreasing or delaying (partially or completely) the need for antiretroviral drug therapy.

ELIGIBILITY:
Inclusion Criteria:

* Prior to any study-related procedures, signed informed consent indicating that they understand the purpose, risks and procedures required for the study and are willing to participate in the study
* Individuals aged 18 to 65 years of age (inclusive) at time of consent
* Documented HIV-1 infection ≥ 6 months prior to Screening 1
* Previous treatment with antiretroviral agents that had a demonstrated suppressive effect (defined as plasma HIV RNA ≤ 50 copies/ml)
* A documented viable ART regimen option, as determined by the Investigator, taking into account prior ART experience and HIV geno/phenotyping analyses
* Not taking antiretroviral therapy for ≥ 6 weeks prior to Screening 1, for one or more of the following reasons:

  i) Concerns over short-term or long-term toxicities associated with antiretroviral agents, or ii) Treatment fatigue from the daily regimen of life-long therapy
* Plasma HIV-1 viral RNA ≥ 5,000 copies/mL and ≤ 100,000 copies/ml at Screening 1 and Screening 2
* CD4+ T lymphocyte count ≥ 500 cells/µl at Screening 1 and Screening 2

Exclusion Criteria:

* Abnormal hematology at Screening 1: Absolute neutrophil count (ANC) < 1.5 x 109/L, Platelet count < 100 x 109/L, Hemoglobin < 10 g/dL
* Abnormal biochemistry at Screening 1: Alanine aminotransferase (ALT) > 2.5 x Upper Limit of Normal (ULN), Total bilirubin > 1.5 x ULN, Serum creatinine > 1.5 x ULN
* Detection of any CXCR4-tropic HIV-1 at Screening 1
* Evidence of co-infection with hepatitis B virus, hepatitis C virus, West Nile Virus, or HTLV-1 as detected at Screening 2
* Evidence of active TB infection determined by positive QuantiFERON®-TB Gold/IGRA test result and clinical confirmation at Screening 2
* ART or other antiretroviral therapy within 6 weeks of Screening 1 or any time during the pre-infusion period
* Documented history of CD4+ T lymphocyte count < 250 cells/µl
* Any previous or current AIDS-defining illnesses (CDC Category C), including AIDS-related dementia, with the exception of Kaposi's sarcoma confined to the skin
* History of malignancy or systemic chemotherapy within the last 5 years (i.e., subjects with prior malignancy must be disease-free for 5 years), except curatively-treated basal cell carcinoma, cutaneous squamous cell carcinoma, or cervical or anal intra-epithelial neoplasia
* History of steroid-dependent asthma in the past 5 years
* History of seizure
* Any clinical history of hematologic diseases including leukemia, myelodysplasia, myeloproliferative disease, thromboembolic disease, sickle cell disorder, thrombocytopenia or leukopenia
* Class II-IV heart failure, according to the New York Heart Association classification
* Inadequate venous access for apheresis, as assessed at Screening 1
* Current or planned systemic immunosuppressive or immunomodulatory medication
* Taking warfarin, aspirin or any medication that is likely to affect platelet function or other aspects of blood coagulation, and unable to safely cease this medication for a period of 1 week prior, during, and 1 week after administration of G-CSF (a total period of 19 days)
* Participation in any study involving any investigational drug or medical device within 30 days prior to Screening 1
* Receipt of a vaccine for HIV-1 or any gene transfer product at any time
* Prior treatment with recombinant G-CSF or busulfan or other stem-cell mobilizing or modulating agent within the previous 12 months
* Known hypersensitivity to busulfan, G-CSF (Neupogen™) or E. coli-derived proteins
* Subjects who will not accept transfusions of blood products
* Pregnant or breast-feeding at any time between Screening 1 and Baseline (infusion)
* History of alcohol or drug abuse within the 12 months prior to Screening 1
* Inability to understand and provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Mitsuyasu, M.D., Principal Investigator — University of California, Los Angeles
Locations (2):
- United States (2):
  - UCLA CARE Center, Los Angeles, California
  - Quest Clinical Research, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 (CSL202 With No Busulfan): Cal-1 modified Hematopoietic stem/progenitor cells (HSPC) and Cal-1 modified CD4+ T lymphocytes (CSL202) without busulfan preconditioning
- Cohort 2 (CSL202 With 1 Busulfan Dose): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes (CSL202), with single 4mg/kg busulfan dose administered as pre-conditioning for transplant
  Busulfan: Intravenous busulfan
- Cohort 3 (CSL202 With 2 Busulfan Doses): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes (CSL202), first busulfan dose = 3mg/kg and second busulfan dose adjusted (total target exposure of 8,000 μmolar/min AUC) administered as pre-conditioning for transplant
  Busulfan: Intravenous busulfan
Period: Overall Study
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Started | 4 | 4 | 5
Completed | 1 | 2 | 1
Not Completed | 3 | 2 | 4
Not completed — Continued to Week 48 but recommenced ART | 3 | 2 | 3
Not completed — Not infused due to manufacturing failure | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 (CSL202 With No Busulfan): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes (CSL202) without busulfan preconditioning
- Cohort 3 (CSL202 With 2 Busulfan Doses): Cal-1 modified HSPC and Cal-1 modified CD4+ T lymphocytes (CSL202), first busulfan dose = 3mg/kg and second busulfan dose adjusted (total target exposure of 8,000 μmolar/min AUC)administered as pre-conditioning for transplant
  Busulfan: Intravenous busulfan
- Total: Total of all reporting groups
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses) | Total
Number analyzed (Participants) | 4 | 4 | 5 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 4 | 5 | 13
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 43.0 (11.7) | 48.5 (12.8) | 46.8 (3.1) | 46.2 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 4 | 4 | 5 | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 1 | 0 | 1
  White | 4 | 3 | 5 | 12
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 4 | 4 | 5 | 13

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Severe and Life-threatening Adverse Events (AEs)
Time Frame: Up to 48 weeks
Population: Safety Population (SP): The safety population includes all enrolled subjects signing informed consent who started the interventional phase of the trial (i.e. CD4+ Apheresis and discontinued subjects who re-commenced ART)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 5
Participants
  Severe | 0 | 4 | 4
  Life-threatening | 0 | 3 | 4

2. Primary Outcome: Number of Participants With Severe or Life-threatening AEs Related to CSL202
Time Frame: Up to 48 weeks
Population: SP
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 5
Participants | 0 | 0 | 1

3. Primary Outcome: Number of Participants With the Presence of Replication-competent Retrovirus
Time Frame: Up to 48 weeks
Population: SP
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 5
Participants | 0 | 0 | 0

4. Primary Outcome: Number of Participants With Predominant Integration Site Analysis
Description: Vector Integration Site Analysis performed only when Cal-1 Marking is >= 1%.
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
Participants | NA — Not done because Cal-1 Marking was <1% at the corresponding time point required | NA — Not done because Cal-1 Marking was <1% at the corresponding time point required | NA — Not done because Cal-1 Marking was <1% at the corresponding time point required

5. Primary Outcome: Mean Cell Dose for CD4+ Cells (Ttn)
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: Number (10^8 cells)
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
Number (10^8 cells) | 16.940 [14.61 to 20.62] | 81.855 [38.94 to 138.68] | 49.553 [20.70 to 79.29]

6. Primary Outcome: Mean Cell Dose for CD34+ Cells (HSPCtn)
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: Number (10^6 cells/kg body weight)
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
Number (10^6 cells/kg body weight) | 2.1 [0.35 to 5.0] | 2.4 [1.0 to 4.0] | 10.6 [7.4 to 12.5]

7. Primary Outcome: Percent Transduction Efficiency of CD4+ Cells (Ttn) and CD34+ Cells (HSPCtn) of Final Cell Product
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: Percent transduction efficiency
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
Percent transduction efficiency
  CD4+ Cells (Ttn) | 41.0 [21.0 to 60.0] | 29.2 [13.0 to 39.0] | 66.8 [39.0 to 84.0]
  CD34+ Cells (HSPCtn) | 58.6 [51.0 to 77.0] | 26.3 [12.0 to 53.0] | 31.3 [21.0 to 49.0]

8. Primary Outcome: Total Area Under the Curve (AUC) for Busulfan
Description: Cohort 3: Total AUC = first dose AUC value + second dose AUC value
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: micromolar*min
Arm/Group | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4
micromolar*min | 6521.5 [5863 to 7259] | 8296.8 [7893 to 8601]

9. Secondary Outcome: Percent Cal-1 Marking in Peripheral Blood
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: percent Cal-1 marking
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
percent Cal-1 marking
  Peak marking | 0.3500 [0.0000 to 1.1600] | 0.7650 [0.6100 to 0.8900] | 3.1200 [0.1800 to 7.4600]
  Week 48 | 0.0000 [0.0000 to 0.0000] | 0.1275 [0.0000 to 0.3800] | 0.1275 [0.0000 to 0.4900]

10. Secondary Outcome: Cal-1 Marking in Gut-associated Lymphoid Tissue (GALT) (10-15 cm)
Description: Samples were collected via endoscopic biopsy from the sigmoid colon: 10-15 cm from the anal margin
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: copies/cell
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
copies/cell
  Peak marking | 0.8121 [0.0 to 2.7054] | 0.0007 [0.0 to 0.0019] | 0.0022 [0.0006 to 0.0060]
  Week 48 | 0.8121 [0.0 to 2.7054] | 0.0004 [0.0 to 0.0010] | 0.0001 [0.0 to 0.0004]

11. Secondary Outcome: Cal-1 Marking in GALT (25-35 cm)
Description: Samples were collected via endoscopic biopsy from the sigmoid colon: 25-35 cm from the anal margin
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: copies/cell
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
copies/cell
  Peak marking | 0.0255 [0.0 to 0.0677] | 0.0003 [0.0 to 0.0011] | 0.0068 [0.0020 to 0.0186]
  Week 48 | 0.0255 [0.0 to 0.0677] | 0.0003 [0.0 to 0.0011] | 0.0055 [0.0 to 0.0186]

12. Secondary Outcome: Cal-1 Marking in Bone Marrow
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: copies/cell
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
copies/cell
  Peak marking | 0.0007 [0.0 to 0.0026] | 0.0539 [0.0005 to 0.2027] | 0.0021 [0.0009 to 0.0030]
  Week 48 | 0.0007 [0.0 to 0.0026] | 0.0015 [0.0005 to 0.0044] | 0.0009 [0.0003 to 0.0025]

13. Secondary Outcome: Cal-1 C46 Expression in Peripheral Blood
Description: C46 relative expression will be analyzed by reverse transcriptase-quantitative polymerase chain reaction (RT-qPCR) and normalized to the expression of β2-microglobulin (β2M) mRNA
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: units of relative expression
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
units of relative expression
  Peak marking | 0.0000 [0.0000 to 0.0000] | 1.0496 [0.0000 to 2.9977] | 2.1701 [0.0000 to 6.4800]
  Week 48 | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000]

14. Secondary Outcome: Cal-1 sh5 Expression in Peripheral Blood
Description: sh5 relative expression will be analyzed by RT-qPCR and normalized to the expression of RNU38B microRNA
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: units of relative expression
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
units of relative expression
  Peak marking | 0.0000 [0.0000 to 0.0000] | 0.2027 [0.0000 to 0.6489] | 1.6933 [0.1930 to 4.6736]
  Week 48 | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000] | 0.0000 [0.0000 to 0.0000]

15. Secondary Outcome: HIV Viral Load at Baseline Screening and Week 48 or at Anti-retroviral Therapy (ART) Re-commencement
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: Log10 (copies/mL)
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
Log10 (copies/mL)
  Baseline screening | 4.59 [4.06 to 4.87] | 4.51 [3.98 to 4.82] | 4.28 [3.45 to 4.62]
  Week 48 or at ART re-commencement | 4.56 [4.00 to 4.93] | 4.70 [3.88 to 4.96] | 4.61 [4.20 to 4.95]

16. Secondary Outcome: CD4+ Count at Baseline Screening and Week 48 or at ART Re-commencement
Time Frame: Up to 48 weeks
Population: SP (1 participant in Cohort 3 withdrew consent and did not receive busulfan or Ttn and HSPCtn)
Measure: Mean (Full Range); unit: CD4+ cells/cubic mm
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 4
CD4+ cells/cubic mm
  Baseline screening | 680.75 [522.5 to 809.5] | 575.13 [537.0 to 677.5] | 668.63 [529.0 to 878.0]
  Week 48 or at ART re-commencement | 553.3 [450 to 759] | 383.5 [274 to 549] | 245.5 [152 to 385]

17. Secondary Outcome: Number of Participants With HIV-1 Tropism Shift
Description: Shift from R5 to X4 or dual/mixed tropism
Time Frame: Up to 48 weeks
Population: SP
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
Number analyzed (Participants) | 4 | 4 | 5
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 48 weeks per participant
Arm/Group | Cohort 1 (CSL202 With No Busulfan) | Cohort 2 (CSL202 With 1 Busulfan Dose) | Cohort 3 (CSL202 With 2 Busulfan Doses)
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/4 | 1/5
Other Adverse Events (participants affected / at risk) | 4/4 | 4/4 | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (CSL202 With No Busulfan) (N=4) | Cohort 2 (CSL202 With 1 Busulfan Dose) (N=4) | Cohort 3 (CSL202 With 2 Busulfan Doses) (N=5)
gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1 (CSL202 With No Busulfan) (N=4) | Cohort 2 (CSL202 With 1 Busulfan Dose) (N=4) | Cohort 3 (CSL202 With 2 Busulfan Doses) (N=5)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 4 (38) | 5 (21)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (19) | 4 (40)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 4 (18) | 3 (4)
Fatigue (General disorders) | 2 (3) | 3 (5) | 3 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (5) | 2 (2)
Nausea (Gastrointestinal disorders) | 0 (0) | 2 (3) | 5 (5)
Diarrhoea (Gastrointestinal disorders) | 1 (3) | 0 (0) | 4 (5)
Upper respiratory tract infection (Infections and infestations) | 3 (5) | 1 (2) | 1 (1)
Chills (General disorders) | 1 (1) | 1 (1) | 3 (3)
Skin odour abnormal (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2) | 0 (0)
Pain (General disorders) | 1 (1) | 1 (1) | 2 (2)
Pyrexia (General disorders) | 1 (1) | 0 (0) | 3 (3)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 3 (3)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 3 (3) | 1 (1)
Headache (Nervous system disorders) | 1 (1) | 1 (1) | 1 (2)
Insomnia (Nervous system disorders) | 1 (1) | 0 (0) | 2 (3)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (4) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0)
Retching (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Toothache (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Asthenia (General disorders) | 0 (0) | 1 (1) | 1 (1)
Malaise (General disorders) | 1 (1) | 1 (1) | 0 (0)
Night Sweats (General disorders) | 0 (0) | 0 (0) | 2 (2)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Acarodermatitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2)
Haematospermia (Reproductive system and breast disorders) | 0 (0) | 1 (2) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Rash vesicular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
ear congestion (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1)
Eye irritation (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Eye pruritus (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Faeces soft (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tongue discolouration (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 1 (1)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gingivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Secondary syphilis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Staphylococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Tinea pedis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 1 (1)
CD4 lymphocytes decreased (Investigations) | 0 (0) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Somnambulism (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Paranasal sinus hypersecretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Tonsillar disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Eosinophilic pustular folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Seborrhoeic dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin erosion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Skin mass (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2015-07-08): https://cdn.clinicaltrials.gov/large-docs/50/NCT01734850/Prot_000.pdf
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/50/NCT01734850/SAP_001.pdf